CLINICAL TRIAL: NCT05839600
Title: An Open-label, Phase I Dose Escalation and Expansion Trial to Investigate Safety and Efficacy of BI 1821736 in Patients With Advanced Solid Tumors
Brief Title: A Study to Find a Suitable Dose of BI 1821736 and Test Whether it Helps People With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1467-0001; 2022-502125-17-00 (Registry Identifier: CTIS (EU)); U1111-1291-2873 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 1821736: Dose escalation cohort (Experimental)
  Interventions: Drug: BI 1821736

INTERVENTIONS:
Drug: BI 1821736 — Solution for infusion

SUMMARY:
This study is open to adults with advanced solid tumours. People with solid tumours for whom previous treatment was not successful or no treatment exists can take part.

The purpose of this study is to find the highest dose of a medicine called BI 1821736 that people with advanced solid tumours can tolerate. BI 1821736 is a type of immunotherapy. It is a special virus that kills cancer cells and helps the immune system fight cancer. In this study, BI 1821736 is given to humans for the first time.

Participants receive BI 1821736 as an infusion into a vein about every 3 weeks for up to 3 months. Study doctors regularly check the participants' health and monitor the tumours. The doctors also take note of any unwanted effects that could have been caused by BI 1821736.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant tumor.
* Advanced, unresectable and/or metastatic or relapsed/refractory solid tumors.
* Has failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patient must have exhausted available treatment options known to prolong survival for their disease.
* Has at least one tumoral lesion which is amenable to biopsy.
* Signed and dated, written informed consent form (ICF) in accordance with ICH-GCP and local legislation obtained prior to any trial-specific procedures, sampling, or analyses that are not part of normal standard of practice care.
* Eastern Cooperative Oncology Group score of 0 or 1.
* Adequate organ function or bone marrow reserve defined as demonstrated at screening by the following laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (≥ 1.5 x 10^3/μL)(≥ 1500/mm^3); haemoglobin ≥ 90 g/L (≥ 9.0 g/dL)(≥ 5.6 mmol/L); platelets ≥ 100 x 10^9/L (≥ 100 x 10^3/μL)(≥ 100 x 10^3/mm^3) without the use of haematopoietic growth factors within 4 weeks of start of trial medication.
  * Creatinine ≤ 1.5 times the upper limit of normal (ULN).
  * Total bilirubin ≤ 1.5 times the ULN, except for patients with Gilbert's syndrome: total bilirubin ≤ 3 times ULN or direct bilirubin ≤ 1.5 times ULN.
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times ULN if no demonstrable liver metastases, or otherwise ≤ 5 x ULN if transaminase elevation is attributable to liver metastases.
  * Partial thromboplastin (PT) / activated partial thromboplastin time (aPTT) <1.5 times ULN unless on a stable dose of an anticoagulant.
  * All toxicities related to previous anti-cancer therapies have resolved to ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 prior to trial treatment administration (except for alopecia and peripheral neuropathy which must be ≤ CTCAE Grade 2 and amenorrhea/menstrual disorders which can be any grade).
* Further inclusion criteria apply

Exclusion Criteria:

* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of study treatment.
* Previous treatment with Vesicular Stomatitis Virus (VSV)-based agents.
* Patients with brain metastases unless they have completed brain radiotherapy and are asymptomatic.
* Radiotherapy within 4 weeks prior to the start of study treatment, except in case of a brief course of palliative radiotherapy (e.g. for analgesic purpose or for lytic lesions at risk of fracture) which can then be completed within two weeks prior to start of study treatment.

Note: No radiation must have been given to any lesions planned to be biopsied within 6 months of start of treatment.

* Prior (within 3 weeks of first dose) or concomitant use of systemic corticosteroids (>10 mg daily prednisone or equivalent).
* Prior (within 3 weeks of first dose or less than 5 half-lives) or concomitant use of a medication or a condition considered a high risk for complications from biopsy as per the Investigator's judgement.
* Prior (within 3 weeks of first dose or less than 5 half-lives) or concomitant use of interferon, immunotherapy agents, or tamoxifen.
* Active infection requiring systemic therapy (antibacterial, antiviral, antiparasitic or antifungal therapy) at the start of treatment in the trial.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLTs) in the Maximum Tolerated Dose (MTD) evaluation period | up to 21 days

SECONDARY OUTCOMES:
Occurrence of DLTs during the on-treatment period | up to 3 months
Occurrence of Adverse Events (AEs) during the on-treatment period | up to 3 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - NEXT Oncology-San Antonio-65273, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto Valenciano de Oncología, Valencia
- Karolinska Universitetssjukhuset Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com